CLINICAL TRIAL: NCT06100809
Title: Personalized Fatigue-Mitigation Lifestyle Coaching (PFMLC) to Improve Performance and Recovery Among Emergency Medicine Residents on Night Shifts
Brief Title: Does Fatigue Coaching Improve Functioning and Fatigue in Resident Night Shifts
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Steven Bird, Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00000500
Record Dates: First submitted 2023-05-10; First posted 2023-10-25 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Fatigue; Shift Work Type Circadian Rhythm Sleep Disorder
Keywords: Fatigue; Shift Work
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Active Comparator): No coaching provided. Nutrional handout only
  Interventions: Behavioral: Nutrition handout
- Intervention (Experimental): Coaching provided. Nutrition handout also provided
  Interventions: Behavioral: Personalized coaching; Behavioral: Nutrition handout

INTERVENTIONS:
Behavioral: Personalized coaching — Personalized fatigue mitigation coaching.
  Arms: Intervention
Behavioral: Nutrition handout — Nutrition handout

SUMMARY:
Emergency Medicine (EM) requires 24/7 staff coverage resulting in healthcare workers' circadian rhythm disruptions that impair clinical and cognitive performance, physical recovery, and contribute to burnout. Multiple well-being surveys continue to highlight EM's challenges with sleep impairment due to the nature of the specialty. Despite evidence that lifestyle strategies effectively optimize performance and recovery, EM residents have variable lifestyle choices to prepare for overnight shifts. This prospective randomized controlled trial will examine whether a pre-shift personalized fatigue-mitigation lifestyle coaching (PFMLC) for EM residents on overnight shifts minimizes the effects of circadian rhythm disruptions on performance and recovery compared to those who receive one-time passive information on lifestyle practices. All participants will receive lifestyle strategy materials on fatigue mitigation to improve performance. Residents' self-reported and biometric data will inform PFMLC in the active arm. Performance and recovery from night shifts will be assessed by changes in sleep, heart rate variability, readiness/recovery, alertness, cognitive performance, and mental health using Fitbit and validated measures.

DETAILED DESCRIPTION:
The investigators will use a block-randomized design utilizing each 28-day scheduling period as a block.

Baseline characteristics and confounding factors such as gender, habitual diet, sleep, and caffeine intake will be collected on the first night of the study. Outcome measures will be assessed at the beginning of the shift and between the hours of 2:00 AM to 5:00 AM when sleep propensity and decreased alertness peak.

Outcome measures include a) Stanford Sleepiness Scale (SSS): which takes about 15 seconds to complete. b) Work Exhaustion (4 questions overall): take 20 seconds to complete. c) electronic psychomotor vigilance test: take 3 minutes to complete. The psychomotor vigilance test is a gamified method to measure both vigilance and reaction time. Done on a phone, a colored block appears on the screen, and when a participant sees the block, the participant taps the screen. Reaction time is measured in milliseconds and the average reaction time over the 3 minutes is calculated by the program and reported to the participant as well as stored in the participant's profile.

Study participants will be required to participate in the study for a total of 18 days. Each study participant will contribute biometric data for 7 days before a string of at least 4 consecutive night shifts, then for another 7 days (for a total of 18 days). A self-care handout containing nutrition tips for fatigue mitigation in night shift workers will be given to all participants at the beginning of the study. A Fitbit device will be provided to all participants to measure biometrics data.

Control: The investigators will not provide personalized coaching and ask the control participants to follow and record their typical nightshift habits. The control participants will participate in the surveys and tests as above. Control participants will receive a daily text message to remind them to do the surveys and tests during their shifts. The investigators will instruct the control participants to make sure their phones are silenced during this time as part of better habits for sleep.

ELIGIBILITY:
Inclusion Criteria:

* emergency medicine resident
* scheduled to work at least 4 overnight consecutive shifts

Exclusion Criteria:

* not willing to wear Fitbit device during the study
* not willing to answer questionnaires
* not willing to receive text messages during the study
* not willing to meet with a lifestyle coach during the study
* not willing t0 download app to their personal smartphone or residency-supplied smartphone

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean of the change in 3 overnight percentage changes (from pre-shift) in mean reaction time | Two time points (beginning and middle of night shifts) on each night for a total of 3 nights]
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  The investigators will compare the mean of the 3 overnight percentage changes from pre to mid-shift between the control and intervention groups for the PVT outcome of mean reaction time reciprocal (lower is desirable).
Mean of the change in 3 overnight percentage changes (from pre-shift) in number of lapses in PVT | Two time points (beginning and middle of night shifts) on each night for a total of 3 nights]
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  The investigators will compare the mean of the 3 overnight percentage changes from pre to mid-shift between the control and intervention groups for the PVT outcome of number of lapses (lower is desirable).
Mean of the change in 3 overnight percentage changes (from pre-shift) in aggregrate PVT score | Two time points (beginning and middle of night shifts) on each night for a total of 3 nights]
  The primary outcome of this study is psychomotor vigilance assessed by the Psychomotor Vigilance Test (PVT) measured by PVT WorkFit iPhone app by Joggle Research by Pulsar. This test takes approximately 3 minutes to complete. The PVT is a widely used objective measure of sustained attention and reaction time, which provides valuable insights into participants' alertness and cognitive performance during different times throughout each of at least 3 consecutive night shifts.
  The investigators will compare the mean of the 3 overnight percentage changes from pre to mid-shift between the control and intervention groups for the PVT outcome of aggregate score (0 worst - 100 best).
Mean of the change in 3 overnight percentage changes (from pre-shift) in Stanford Sleepiness Scale | Two time points (beginning and middle of night shifts) on each night for a total of 3 nights]
  The Sleepiness Symptom Scale (SSS) is a validated subjective measure of sleepiness frequently used for research and clinical purposes. It evaluates sleepiness at specific moments in time using a single-item scale. Respondents select one of seven statements to indicate their level of perceived sleepiness. Score Range: The scale score ranges from 1 to 7, reflecting the varying degrees of sleepiness experienced by respondents. This test takes approximately 15 seconds to complete.
  Directionality: Higher scores on the SSS represent higher perceived sleepiness, while lower scores indicate increased alertness and desirable.
  The investigators will compare the mean of the 3 overnight percentage changes from pre to mid-shift between the control and intervention groups.
Mean of the change 3 overnight percentage changes (from pre-shift) in Noordsy-Dahle Subjective Experience Scale (NDSE) Modified version of Noordsy-Dahle Subjective Experience Scale (NDSE) for healthy adults includes 8 sub-domains: | Two time points (beginning and middle of night shifts) on each night for a total of 3 nights]
  Global well-being: Delighted 1 to Terrible 7, Lower score better Anxiety: None 1 to Extreme 7, Lower score better Depression: None 1 to Extreme 7, Lower score better Energy: Tired 1 to Energized 7, Higher score better Motivation: None 1 to Strong 7, Higher score better Clarity of thought: Clouded 1 to Totally Clear 7, Higher score better Concentration: Poor 1 to Excellent 7, Higher score better Social interest: Alone 1 to With Others 7, Higher score better This test takes approximately 90 seconds to complete.We will compare the mean of the 3 overnight percentage changes from pre to mid-shift between the control and intervention groups

SECONDARY OUTCOMES:
Mean of total hours of sleep | 1 week of baseline, during the 1 week of night shifts, and for 1 week after the night shifts
  Total sleep hours per 24-hour period during a baseline week, the period of night shifts, and a recovery week using FitBit Versa 4, between the two groups will be compared.
Mean of heart rate variability | 1 week of baseline, during the week of night shifts, and for 1 week after the night shifts
  Heart rate variability per 24-hour period during a baseline week, the period of night shifts, and a recovery week using Fitbit Versa 4, between the two groups will be compared.

OTHER OUTCOMES:
Percentage change from baseline in NIH PROMIS Short Form Sleep-Related Impairment | 1 week of baseline, during the week of night shifts, and for 1 week after the night shifts
  The NIH PROMIS Short Form Sleep-Related Impairment Scale is included as an exploratory outcome measure in this study. The Sleep-Related Impairment is designed to assess the impact of sleep-related impairment on various aspects of daily functioning and overall quality of life. Higher scores indicate greater sleep-related impairment. The NIH PROMIS takes about 1 minute to complete and will be measured at the beginning of the study and at the end of the study. The investigators will compare the percentage change from baseline between the two groups.
Percentage change from baseline in Task Load Index | 1 week of baseline, during the week of night shifts, and for 1 week after the night shifts
  The National Aeronautics and Space Administration\ (NASA) Task Load Index (TLX) is included as an exploratory outcome measure in this study. The TLX is used to measure cognitive load. Lower scores are more desirable. The TLX takes about 1 minute to complete and will be measured at the beginning of the study and at the end of the study. The investigators will compare the percentage change from baseline between the two groups.

CONTACTS AND LOCATIONS:
Locations (1):
- UMassMemorial Health Care, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No